CLINICAL TRIAL: NCT03515057
Title: Screening for Atrial Fibrillation in an Ambulatory Clinic Population: The VITAL-AF Study
Brief Title: Screening for Atrial Fibrillation Among Older Patients in Primary Care Clinics
Acronym: VITAL-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Steven A Lubitz, Cardiac Electrophysiologist, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CV185-581
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial Fibrillation Spot-Check (Experimental): For eligible patients from primary care clinics randomly selected for the Atrial Fibrillation Spot-Check arm, practice medical assistants will screen assenting patients for undiagnosed AF during regularly scheduled office visits using a single-lead handheld electrocardiogram (ECG). Single-lead handheld electrocardiogram readings detecting AF will be confirmed during the same office visit with a standard 12-lead ECG at the discretion of the primary care physician. If AF is detected, the patient's PCP will be able to address the condition with them during the clinic visit and initiate appropriate follow-up to manage the AF.
  Interventions: Diagnostic Test: Single lead handheld electrocardiogram
- Usual Care (No Intervention): For eligible patients from primary care clinics randomly selected for the Usual Care arm, they will receive standard care during outpatient visits without change.

INTERVENTIONS:
Diagnostic Test: Single lead handheld electrocardiogram — Screening for atrial fibrillation during outpatient primary care office visits among patients 65 years and older
  Other Names: AliveCor KardiaMobile EKG Monitor
  Arms: Atrial Fibrillation Spot-Check

SUMMARY:
The overall goal of this study is to assess the effectiveness of screening for undiagnosed atrial fibrillation (AF) using simple, efficient, and portable electronic health and mobile technologies in a healthcare system. The investigators propose to perform population-based screening for undiagnosed AF as part of usual care in patients ≥ 65 years when their vital signs are checked (spot-check) at scheduled outpatient visits in adult Massachusetts General Hospital (MGH) primary care clinics. Patients will receive routine care by their primary care provider (PCP) based upon the results of the screening during the visit.

The investigators hypothesize that rates of AF detection among individuals ≥ 65 years in the MGH primary care network will be greater among patients in clinics assigned to the spot-check arm compared to patients in clinics assigned to the usual care arm of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older
* Presenting for an outpatient clinic appointment at a participating clinic
* Visit with a physician, nurse practitioner, or physician's assistant

Exclusion Criteria:

* Have a primary care physician outside of the network
* Do not visit their primary care practice during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35308 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Incident AF during the study period | 12-months
  The numerator of the outcome is the number of eligible patients with newly diagnosed AF during the study period. The eligible study population comprising the denominator will be assessed in two ways: (1) the whole population, defined as all patients aged 65 years and older presenting for an outpatient clinic appointment with a participating physician, nurse practitioner, or physician assistant at a study clinic during the enrollment period, and (2) the whole population excluding patients with an AF diagnosis prior to outcome assessment (prevalent AF).

SECONDARY OUTCOMES:
Incident AF associated with a primary care encounter during the study period | 12-months
  The numerator of the outcome will be the number of eligible patients with newly diagnosed AF associated with a primary care visit. Similar to the primary outcome, the denominator will be assessed in two ways: (1) the whole population, and (2) the whole population excluding prevalent AF.
New oral anticoagulation prescription during the study period | 12-months
  The numerator of the outcome will be the number of eligible individuals with a new oral anticoagulation prescription during the study period. The eligible study population comprising the denominator will be assessed in three ways: (1) the whole population, (2) patients with a new AF diagnosis (incident AF), and (3) patients with prevalent AF.
Continued prescription of anticoagulation at 12 months among those started on anticoagulation during the study period | 12-months following initial prescription of anticoagulation (ie, up to 24 months after study start)
  The numerator will be the number of individuals with a refill or prescription of an alternative anticoagulant in the subsequent 12 months after the day of new anticoagulant prescription. The eligible study population comprising the denominator will include individuals who are started on OAC during the study period. The denominator will be assessed in three ways: (1) whole population, (2) incident AF and (3) prevalent AF.
New ischemic stroke within 24-months of the study start | 24-months
  The numerator of the outcome is the number of patients sustaining ischemic stroke within 24 months of the study start. The eligible study population comprising the denominator will be assessed in two ways: (1) whole population, and (2) patients with an AF diagnosis (prevalent AF or incident AF prior to the outcome).
Major hemorrhage within 24-months of the study start | 24-months
  The numerator of the outcome is the number of patients sustaining a major hemorrhagic event within 24 months of the study start. The eligible study population comprising the denominator will be assessed in two ways: (1) whole population, and (2) patients with an AF diagnosis (prevalent AF or incident AF prior to the outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lubitz, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khurshid S, Friedman SF, Al-Alusi MA, Kany S, Sommers T, Anderson CD, Ho JE, McManus DD, Borowsky LH, Ashburner JM, Lubitz SA, Atlas SJ, Maddah M, Singer DE, Ellinor PT. Artificial intelligence-enabled analysis of handheld single-lead electrocardiograms to predict incident atrial fibrillation: an analysis of the VITAL-AF randomized trial. NPJ Digit Med. 2025 Nov 26;8(1):776. doi: 10.1038/s41746-025-02164-2. PMID 41299008
- [Derived] Atlas SJ, Ashburner JM, Chang Y, Borowsky LH, Ellinor PT, McManus DD, Lubitz SA, Singer DE. Screening for undiagnosed atrial fibrillation using a single-lead electrocardiogram at primary care visits: patient uptake and practitioner perspectives from the VITAL-AF trial. BMC Prim Care. 2023 Jun 30;24(1):135. doi: 10.1186/s12875-023-02087-5. PMID 37391738
- [Derived] Lubitz SA, Atlas SJ, Ashburner JM, Lipsanopoulos ATT, Borowsky LH, Guan W, Khurshid S, Ellinor PT, Chang Y, McManus DD, Singer DE. Screening for Atrial Fibrillation in Older Adults at Primary Care Visits: VITAL-AF Randomized Controlled Trial. Circulation. 2022 Mar 29;145(13):946-954. doi: 10.1161/CIRCULATIONAHA.121.057014. Epub 2022 Mar 2. PMID 35232217
- [Derived] Ashburner JM, Atlas SJ, McManus DD, Chang Y, Trisini Lipsanopoulos AT, Borowsky LH, Guan W, He W, Ellinor PT, Singer DE, Lubitz SA. Design and rationale of a pragmatic trial integrating routine screening for atrial fibrillation at primary care visits: The VITAL-AF trial. Am Heart J. 2019 Sep;215:147-156. doi: 10.1016/j.ahj.2019.06.011. Epub 2019 Jun 22. PMID 31326680